CLINICAL TRIAL: NCT05978167
Title: Targeting Neural, Behavioral and Pharmacological Mechanisms of Drug Memories in Drug Addiction With Methylphenidate
Brief Title: Targeting Drug Memories With Methylphenidate
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rita Goldstein, Chief of Research, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 20-2707; R21DA054281 (NIH)
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorder; Cocaine Use Disorder
MeSH Terms: conditions — Substance-Related Disorders | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylphenidate then Placebo (Experimental): 20 mg of methylphenidate then matching placebo pill.
  Interventions: Drug: Methylphenidate; Behavioral: Memory reconsolidation; Drug: Placebo
- Placebo then Methylphenidate (Placebo Comparator): Matching placebo pill then 20 mg of methylphenidate.
  Interventions: Drug: Methylphenidate; Behavioral: Memory reconsolidation; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Oral administration of 20 mg Methylphenidate
Behavioral: Memory reconsolidation — Retrieval of drug-cue memories before extinction.
Drug: Placebo — Matching placebo pill

SUMMARY:
This study aims to identify the neural, behavioral, and pharmacological mechanisms promoting diminished expression of drug-related memories in human drug addiction. In this fMRI study with a within-subjects placebo-controlled double-blind cross-over design, oral methylphenidate (20 mg) or placebo will be administered to individuals with cocaine use disorders (CUD) to peak during the retrieval of a drug-cue memory before extinction; in addition to fMRI activations, skin conductance responses (SCR, acquired simultaneously) will serve as the psychophysiological indicators of memory modification. Assessments of interference with the return of drug-cue memories via SCR and craving will be conducted the day following MRI. This pharmocologically-enhanced behavioral approach to decreasing drug memories and craving in iCUD could ultimately be used to develop effective cue-exposure therapies for drug addiction. Procedures include MRI, blood draw, questionnaires and interviews, skin conductance response measures, and behavioral tasks.

DETAILED DESCRIPTION:
Cue-exposure therapy has not proven efficacious in reducing relapse in drug addiction, illuminating the need for alternative strategies. Here researchers will test the neural correlates of two strategies, encompassing behavioral and pharmacological approaches, aimed to interfere with the return of drug memories in individuals with cocaine use disorders. Results may pave the way towards enhancing the efficacy of cue-exposure therapy in reducing cue-induced craving and relapse in drug addiction (generalizable across drugs of abuse/behavioral addictions).

ELIGIBILITY:
Inclusion criteria:

* Ability to understand and give informed consent
* Males and females, 18-65 years of age
* DSM-V diagnosis for CUD or otherwise problematic cocaine use as clinically determined

Exclusion criteria:

* DSM-5 diagnosis for schizophrenia or developmental disorder (e.g., autism)
* Head trauma with loss of consciousness
* History of neurological disease of central origin including seizures
* Cardiovascular disease including high blood pressure and/or other medical conditions, including metabolic, endocrinological, oncological or autoimmune diseases, and infectious diseases including Hepatitis B and C or HIV/AIDS
* Metal implants or other MR contraindications

Ages: 26 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
fMRI blood-oxygenation level dependent (BOLD) signal | Day 1
  fMRI blood-oxygenation level dependent (BOLD) signal deactivation in the ventromedial prefrontal cortex in response to retrieval of drug-cue memory.
fMRI blood-oxygenation level dependent (BOLD) signal | Day 7
  fMRI blood-oxygenation level dependent (BOLD) signal deactivation in the ventromedial prefrontal cortex in response to retrieval of drug-cue memory.

SECONDARY OUTCOMES:
Skin Conductance Responses (SCR) | 24 hours after each neuroimaging session
  Measure of changes to skin conductance responses in response to retrieval of drug-cue memory. The conductance is measured by placing two electrodes on the fingers and passing a small, 0.5 V electric charge between the two points. An increase in the skin conductance response (SCR) reflects heightened arousal in response to the drug-cue memory, changes in which are monitored following exposure to the drug cues.
Craving | 24 hours after each neuroimaging session
  Measure of changes to craving in response to retrieval of drug-cue memory. Self-reported cue-induced craving in response to drug cues will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Z Goldstein, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to rita.goldstein@mssm.edu. To gain access, data requestors will need to sign a data access agreement.